CLINICAL TRIAL: NCT03253354
Title: Exploring Novel Neurostimulation Based Therapies for Swallowing Impairments in Parkinson's Disease
Brief Title: Neurostimulation for Dysphagia in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Prof Shaheen Hamdy PhD FRCP, Professor of Neurogastroenterology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS: 200591
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Dysphagia; Parkinson Disease; Swallowing Disorder.Other Specified; Brain Diseases
MeSH Terms: conditions — Deglutition Disorders; Parkinson Disease; Brain Diseases | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: 4 arm randomised single dose study
Who Masked: Participant
Masking Description: Patient blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pharyngeal stimulation (Active Comparator): Pharyngeal stimulation given at 5Hz for 10 minutes
  Interventions: Device: repetitive magnetic stimulation
- repetitive magnetic stimulation (1Hz) (Active Comparator): repetitive transcranial magnetic stimulation at 1Hz applied for 600 pulses
  Interventions: Device: repetitive magnetic stimulation
- repetitive magnetic stimulation (5Hz) (Active Comparator): repetitive transcranial magnetic stimulation at 5Hz applied for 600 pulses
  Interventions: Device: repetitive magnetic stimulation
- Sham treatment (Sham Comparator): Sham repetitive transcranial magnetic stimulation using the coil tilt technique
  Interventions: Device: repetitive magnetic stimulation

INTERVENTIONS:
Device: repetitive magnetic stimulation — Neurostimulation
  Other Names: pharyngeal stimulation

SUMMARY:
This study will explore the effects of 3 different neurostimulation methods on swallowing function in patients with dysphagia secondary to Parkinson's Disease

DETAILED DESCRIPTION:
The aim of this study is to assess 3 novel neuromodulation approaches - namely, pharyngeal stimulation, high frequency (5Hz) repetitive transcranial magnetic stimulation and low frequency (1Hz) repetitive transcranial magnetic stimulation on swallowing function in patients with dysphagia after Parkinson's Disease. A total of 66 patients are planned to be recruited, randomised to one of the 3 technologies or a sham treatment. A single treatment will be given and the effects will be assessed with a barium exam called videofluoroscopy within the 1st hour after the treatment. In addition, some measures of brain function will be recorded, before and after the treatments using single pulse transcranial magnetic stimulation.

ELIGIBILITY:
Inclusion Criteria:

Confirmed Parkinson's Disease with dysphagia

Exclusion Criteria:

Contraindications to magnetic stimulation, such as pacemakers, significant neuroleptic medications, pregnancy Other causes for dysphagia Unable to give informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Videofluoroscopy | 1 hour
  Changes in penetration aspiration scale

SECONDARY OUTCOMES:
Brain excitability | Immediately after, 30 and 60 minutes
  Measures of brain function to single pulse TMS

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Hamdy, PhD FRCP, Principal Investigator — University of Manchester
Locations (1):
- Salford Royal Hospital, Salford, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized swallowing physiology data